CLINICAL TRIAL: NCT03330912
Title: The Influence of Seat Height on Hemiplegic-pattern Propulsion of Manual Wheelchairs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lee Kirby (Other)
Responsible Party: Sponsor-Investigator, Lee Kirby, Staff Physician, Rehabilitation Medicine, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1022716
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Wheelchairs; Hemiplegia
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Intervention Model Description: Single subject - participants will be compared to themselves. STROBE guidelines will be followed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Seat Height Intervention (Experimental): Randomly assigned 5 wheelchair seat heights ranging from very low (2" below) to very high (2" above) the lower leg length of the participant.
  Interventions: Device: Neutral seat height; Device: Very low seat height; Device: Low seat height; Device: Very high seat height; Device: High seat height

INTERVENTIONS:
Device: Neutral seat height — Seat height set relative to participant's leg length with neutral set at the measured lower leg length
Device: Very low seat height — Seat height set relative to participant's leg length, 2" below the measured lower leg length
Device: Low seat height — Seat height set relative to participant's leg length, 1" below the measured lower leg length
Device: Very high seat height — Seat height set relative to participant's leg length, 2" above the measured lower leg length
Device: High seat height — Seat height set relative to participant's leg length, 1" above the measured lower leg length

SUMMARY:
This study evaluates the effect of seat height on hemiplegic-pattern wheelchair propulsion. Each subject will act as their own control and measures will be obtained in a one sixty minute session. Five seat heights relative to the subject's leg length will be measured in a random order to see the effect on forward and backwards wheelchair propulsion.

DETAILED DESCRIPTION:
Many people who have suffered a stroke require a wheelchair for mobility. Hemiplegia is a common result of stroke.Many people with hemiplegia propel themselves using their sound-side arms and legs ("hemiplegic-pattern propulsion") in manual wheelchairs.Often people using this pattern are prescribed wheelchairs with a reduced seat height to facilitate foot propulsion. Despite the seeming obviousness of the need to lower the seat height for people who use foot propulsion,there is little available evidence to help establish optimal wheelchair seat height. The study objective is to test the hypothesis that there is an optimum wheelchair seat height (expressed as a percentage of the lower leg length) for hemiplegic-pattern wheelchair propulsion. The investigators expect that the optimum seat height will be lower than that usually used for wheelchairs that are hand-propelled.

A single-subject design with able-bodied participants will be used to investigate 5 randomized seat heights. The 5 seat heights will be set relative to the subjects leg length at a single 60 minute data collection session All measures will be obtained during one session. The optimal seat height will be chosen based on wheelchair propulsion speed, push frequency and effectiveness over 10m going forward on smooth surface, and 5m going backwards over a soft surface.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate
* is right-hand dominant (to simplify wheelchair and laboratory set-up)
* has a subjective unshod height of ≤ 183 cm (6'0")
* is able to be comfortably seated in the manual wheelchair used for the study
* is 18 years of age or older, is alert and cooperative
* is competent to provide informed consent
* is able to communicate in English
* does not have an unstable medical condition

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
speed (m/s) | same day measure obtained immediately after seat adjustment, approximately 10 minutes
  wheelchair propulsion speed over 10 m forward and 5 m backward
push frequency (cycles per second) | same day measure obtained immediately after seat adjustment, approximately 10 minutes
  number of foot cycles completed over the 10 m forward and 5 m backward
Propulsion effectiveness | same day measure obtained immediately after seat adjustment, approximately 10 minutes
  distance travelled per foot propulsion cycle

SECONDARY OUTCOMES:
forward propulsion wheelchair skills test score | same day measure obtained immediately after seat adjustment, approximately 10 minutes
  fail, pass with difficulty or pass for wheeling forward 10 m
propulsion difficulty questionnaire | same day measure obtained immediately after seat adjustment, approximately 10 minutes
  Investigator developed questionnaire asking how difficult it was to perform the propulsion test. The participant will self-report his/her level of difficulty for this skill using a five-point Likert scale (1 =very easy, 2=somewhat easy, 3=neither easy nor difficult, 4= somewhat difficult and 5=very difficult). A single number will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Kirby, MD, Principal Investigator — Nova Scotia Health Authority, Dalhousie University
Locations (1):
- Nova Scotia Rehabilitation and Arthritis Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heinrichs ND, Kirby RL, Smith C, Russell KFJ, Theriault CJ, Doucette SP. Effect of seat height on manual wheelchair foot propulsion, a repeated-measures crossover study: part 1 - wheeling forward on a smooth level surface. Disabil Rehabil Assist Technol. 2021 Nov;16(8):831-839. doi: 10.1080/17483107.2020.1741036. Epub 2020 Apr 2. PMID 32238086
- [Background] Heinrichs ND, Kirby RL, Smith C, Russell KFJ, Theriault CJ, Doucette SP. Effect of seat height on manual wheelchair foot propulsion, a repeated-measures crossover study: part 2 - wheeling backward on a soft surface. Disabil Rehabil Assist Technol. 2022 Apr;17(3):325-330. doi: 10.1080/17483107.2020.1782490. Epub 2020 Jun 27. PMID 32594783